CLINICAL TRIAL: NCT07284862
Title: A Cross-sectional Study on the Association of Peptidoglycan Fragments Derived From Gut Microbiota With Alcohol Liver Disease
Status: Completed | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZhujingGS
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Alcohol-associated Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALD-related cirrhosis: This cohort consists of patients with alcohol-related liver cirrhosis, diagnosed based on clinical-pathological assessment with confirmation by two hepatologists. All patients had chronic liver disease for ≥6 months with an established etiology (primarily alcohol-related, defined as >2 oz/day ethanol for men or >1 oz/day for women for >10 years). Key exclusions include recent (within 1 month) use of antibiotics/probiotics/PPIs, recent (within 6 months) gastrointestinal procedures, and presence of uncontrolled infection or hypertension.
  Interventions: Other: An observational, non-interventional study design.
- health: This cohort consists of age- and sex-matched healthy controls recruited from a Health Checkup Center, with no clinically diagnosed chronic diseases.
  Interventions: Other: An observational, non-interventional study design.

INTERVENTIONS:
Other: An observational, non-interventional study design. — An observational, non-interventional study design.

SUMMARY:
alcohol-associated liver disease (ALD) is a leading cause of cirrhosis, yet the role of gut microbiota-derived peptidoglycan (PG) metabolites in liver injury remains unclear. This study aimed to elucidate the role of microbial DL-endopeptidases, which generate NOD2 ligands, in modulating alcohol-induced liver injury.Participants will provide stool samples.

ELIGIBILITY:
Inclusion Criteria:

(1) patients diagnosed with liver cirrhosis based on clinical-pathologic features including liver history and endoscopic or radiologic findings (the presence of clinical cirrhosis was adjudicated in a blinded fashion by two separate hepatology experts; to be included, both experts were required to agree on the presence of clinical cirrhosis) and (2) all patients with chronic liver disease were required to have evidence of clinical liver disease for at least 6 months and were required to have an identifiable etiology of liver disease, including alcohol-related liver diseases (based on a history of alcohol use disorder or a past history of alcohol consumption of greater than 2 ounces of ethanol per day for men or 1 ounce of ethanol per day for women (for greater than 10 years) with no other cause of liver disease identified), NAFLDs, viral hepatitis B or C (detected by HCV RNA or HBV DNA measurement) or autoimmune liver disease (based on international autoimmune scoring criteria).

Exclusion Criteria:

(1) individuals treated with antibiotics, probiotics or proton pump inhibitors within 1 month before sample collection; (2) any participant undergoing a gastrointestinal surgical procedure or colonoscopy within 6 months before sample collection; (3) any individual with uncontrolled infection; and (4) individuals with uncontrolled systolic blood pressure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Meet eligibility criteria
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Fecal NOD2-stimulating activity, measured using a HEK-Blue-hNOD2 reporter cell assay. | Baseline (pre-treatment)
  To explore the potential of peptidoglycan fragments as screening or diagnostic biomarkers for alcohol-related liver disease.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong He, xiaolong, Study Director — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China